CLINICAL TRIAL: NCT04146779
Title: Feasibility Study of a Yoga Intervention in Head and Neck Cancer Patients Undergoing Concurrent Chemo-Radiation
Brief Title: Yoga Intervention in Head and Neck Cancer Patients Undergoing Concurrent Chemo-Radiation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19
Sponsor: Vanderbilt-Ingram Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Barbara Murphy, MD, Sponsor Investigator, Vanderbilt-Ingram Cancer Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: VICC SUPP 18154
Record Dates: First submitted 2019-10-29; First posted 2019-10-31 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Posture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video and Written Yoga Instruction (Experimental): Videos and written instructions on Hatha yoga will be provided
  Interventions: Behavioral: Yoga Video; Behavioral: Posture and Strengthening Video; Behavioral: Relaxation Video; Behavioral: Breath Work Video; Behavioral: Satisfaction Survey; Behavioral: Written Yoga Instructions
- Video, Written Yoga Instruction Plus Guided Yoga Sessions (Experimental): Videos and written instructions on Hatha yoga and instructor guided session on Hatha yoga will be provided
  Interventions: Behavioral: Yoga Video; Behavioral: Posture and Strengthening Video; Behavioral: Relaxation Video; Behavioral: Breath Work Video; Behavioral: Satisfaction Survey; Behavioral: Guided Yoga Session; Behavioral: Written Yoga Instructions

INTERVENTIONS:
Behavioral: Yoga Video — A guided practice that includes gentle stretching of the jaw, neck and shoulders. It lasts approximately 25 minutes.
Behavioral: Posture and Strengthening Video — The strengthening video directs patients through a sequence of isometric exercises to strengthen neck, shoulder and core muscles that are critical for good posture and musculoskeletal integrity. The patient may opt to do the strengthening exercises standing, sitting or with their back on the floor depending on their strength. The video lasts 20 minutes.
Behavioral: Relaxation Video — The relaxation video uses meditative techniques to quiet and calm the mind. The video lasts 15 minutes
Behavioral: Breath Work Video — The breath work video will guide patients through a series of abdominal and chest breathing exercises. The video lasts 15 minutes.
Behavioral: Satisfaction Survey — Participants will complete a questionnaire addressing satisfaction with the yoga program.
Behavioral: Guided Yoga Session — Instructor guided yoga session twice a week
  Arms: Video, Written Yoga Instruction Plus Guided Yoga Sessions
Behavioral: Written Yoga Instructions — Introduction to Yoga and Yoga poses

SUMMARY:
This is a randomized prospective pilot study assessing the safety and feasibility of two yoga interventions in head and neck cancer patients undergoing primary or adjuvant radiation with or without concurrent chemotherapy

DETAILED DESCRIPTION:
Primary Objective:

- To assess the safety and feasibility of Hatha yoga in head and neck cancer patients undergoing treatment with primary or adjuvant radiation with or without chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced, non-metastatic, histologically confirmed malignancy involving the head and neck region

  o Larynx, pharynx, oral cavity, salivary gland, paranasal sinuses and unknown primary
* Age greater or equal to 21 years of age
* Planned for either definitive or adjuvant radiation therapy with or without chemotherapy

  o Patients may have received induction chemotherapy or primary surgical resection prior to proceeding to radiation therapy
* Ability to understand English
* Daily access to the internet
* Willing and able to sign informed consent
* Willing and able to participate in yoga sessions as outlined in the study protocol

Exclusion criteria:

* Prior head and neck cancer radiation
* Patients who in the opinion of the treating physician are physically, medically or psychologically impaired to the point that participation is not deemed appropriate or feasible

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-10-06 (Actual); Study Completion 2020-10-06 (Actual)

PRIMARY OUTCOMES:
Safety of Hatha yoga | Approximately 8 weeks
  Number of adverse events as graded by CTCAE 4.0
Feasibility of Hatha yoga | Approximately 8 weeks
  At least 50% of patients will need to moderately compliant to be feasible (Compliance will be defined as:Fully Compliant: Participation in at least 1 yoga activity on at least 70% of days on study; Moderately Compliant: Participation in at least 1 yoga activity on at least 40% of days on study;Noncompliant: Participation on less than 40% of days on study)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Murphy, MD, Principal Investigator — Vanderbilt-Ingram Cancer Center
Locations (1):
- Vanderbilt-Ingram Cancer Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No